CLINICAL TRIAL: NCT00045864
Title: Proleukin in Combination With Rituxan in Patients With Intermediate and High-Grade Non-Hodgkin's Lymphoma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiron Corporation (Industry)
Purpose: Treatment
Other Study IDs: IL2NHL05
Record Dates: First submitted 2002-09-12; First posted 2002-09-16 (Estimated); Last update posted 2006-02-06 (Estimated); Status verified 2006-02

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Intermediate and High-Grade Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — aldesleukin; Rituximab

INTERVENTIONS:
Drug: Recombinant Human Interleukin-2 and Rituximab

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of combination therapy with Proleukin and Rituxan on patients with intermediate-and high- grade Non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion:

* Diagnosis: CD20+ B-cell non-Hodgkin's lymphoma (NHL) classified as intermediate- or high-grade according to the Working Formulation, subtypes D to H. Must have measureable progressive or refractory disease after no more than three prior chemotherapy regimens.

Exclusion:

* Clinically significant cardiac dysfunction, or a history of myocardial infarction or heart failure within 6 months of first study treatment
* Clinically significant pulmonary dysfunction.
* Liver disease (note hepatitis C seropositive subjects may be enrolled if they have no active disease as demonstrated by undetectable HCV viral loads, biopsy showing no active disease, and/or history of normal transaminases on at least three different dates within one year of first study treatment).
* Symptomatic thyroid disease requiring medical intervention other than replacement treatment for hypothyroidism.
* History of autoimmune disease.
* History of positive serology for human immunodeficiency virus (HIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - ACRC/Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Hoag Cancer Center, Newport Beach, California
  - UC Davis Cancer Center, Sacramento, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Stanford University Medical Center, Stanford, California
  - California Cancer Medical Center, West Covina, California
  - Georgetown University Medical Center, Lombardi Cancer Center, Washington D.C., District of Columbia
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Division of Hematology/Oncology, University of Miami School of Medicine, Miami, Florida
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Rush Cancer Institute, Chicago, Illinois
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Cancer Care Center, Bloomington, Indiana
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Louisiana Health Sciences Center, Department of Medicine, Hematology/Oncology, Shreveport, Louisiana
  - Kansas City Oncology and Hematology Group, Kansas City, Missouri
  - Arch Medical Group, LLC, St Louis, Missouri
  - Dartmouth-Hitchcock-Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Our Lady of Mercy Medical Center, Comprehensive Cancer Center, The Bronx, New York
  - East Carolina University School of Medicine/ Division of Hematology/Oncology, Greenville, North Carolina
  - Roger Maris Health System, Fargo, North Dakota
  - Gabrail Cancer Center, Canton, Ohio
  - Oncology Hematology Care Inc., Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Hematology /Oncology Consultants Inc., Columbus, Ohio
  - Oregon Heath and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Germantown Cancer Center, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cancer Specialists of South Texas, P.A., Corpus Christi, Texas
  - Virginia Cancer Institute, Richmond, Virginia